CLINICAL TRIAL: NCT05386966
Title: Medicolegal Aspects of Head Trauma in Sohag University Hospitals
Brief Title: Medicolegal Aspects of Head Trauma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Naglaa Gaber Ahmed, Demonstrator of Forensic Medicine & Clinical Toxicology Faculty of Medicine_ SohagUniversity, Sohag University
Other Study IDs: Soh-Med-22-05-02
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Head Trauma
MeSH Terms: conditions — Craniocerebral Trauma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — Patient demographic data ( age, gender, residence , work ,Level of education) .Detailed history about the trauma (type, site , manner , mechanism of injury , actual cause of assault , post traumatic period till arrival to hospital ) .Clinical assessment ( Rapid neurological assessment , assesment of Scalp injury ,Presence of other body trauma ,Degree of severity of head injury according to GCS , Radiological finding. Treatment (Conservative or operative intervention ) .Follow up and outcome at the time of discharge by using the GOS .Expected time for healing (<20 day or >20 day ).Expectance for permanent infirmity

SUMMARY:
Trauma is a critical global health problem. It represents the fifth leading cause of significant disability and is one of the most common causes of mortality in youth and adulthood, as one in 10 deaths worldwide occurred due to trauma.

The head is preferred target for criminal acts and is a favorite place for various pathological lesions .Traumatic head injury (THI)is one of the prevalent causes of global death and disability. lately, head injury (HI) cases have increased in both developed and developing nations. Therefore, it is of great value to evaluate the clinical and pathological features of head injury .

Every injury that results in harm to the scalp, skull or brain can be sort out as a HI which can be caused by traffic mishap, falls, sports and gunshot wounds. Vehicle accidents are one of the most prevalence causes of THI as they are deemed to be one of the main causes of fatality due to road-traffic accidents (RTA) .Among different type of the RTA, motorcycle accidents holds the number one cause of accident in most of the country .

Skull fracture and hemorrhage are common association, which may be present with head trauma and affect the outcome of the case.The skull fractures, especially by blunt force offer varying diagnostic and medico- legal problems to the medical jurists as well as to the clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of head trauma

Exclusion Criteria:

* Patients with deficient data i.e. escaped, discharged on demand before period of follow up

Min Age: 1 Day | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosed cases of head trauma at Department of Neurosurgery
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The aim of the current study is to assess and describe the change in the medicolegal aspects of traumatic head injuries in sohag university hospital | 1year
  Expected time for healing and expectance for permanent infirmity

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chelly H, Bahloul M, Ammar R, Dhouib A, Mahfoudh KB, Boudawara MZ, Chakroun O, Chabchoub I, Chaari A, Bouaziz M. Clinical characteristics and prognosis of traumatic head injury following road traffic accidents admitted in ICU "analysis of 694 cases". Eur J Trauma Emerg Surg. 2019 Apr;45(2):245-253. doi: 10.1007/s00068-017-0885-4. Epub 2017 Dec 12. PMID 29234838
- [Background] Wang J, Han F, Zhao Q, Xia B, Dai J, Wang Q, Huang S, Le C, Li Z, Liu J, Yang M, Wan C, Wang J. Clinicopathological Characteristics of Traumatic Head Injury in Juvenile, Middle-Aged and Elderly Individuals. Med Sci Monit. 2018 May 18;24:3256-3264. doi: 10.12659/MSM.908728. PMID 29773781
- [Background] Pearn ML, Niesman IR, Egawa J, Sawada A, Almenar-Queralt A, Shah SB, Duckworth JL, Head BP. Pathophysiology Associated with Traumatic Brain Injury: Current Treatments and Potential Novel Therapeutics. Cell Mol Neurobiol. 2017 May;37(4):571-585. doi: 10.1007/s10571-016-0400-1. Epub 2016 Jul 6. PMID 27383839